CLINICAL TRIAL: NCT04703049
Title: The Effect of Whole Blood Viscosity on Contrast-Induced Nephropathy Development in Patients Undergoing Elective Percutaneous Coronary Intervention
Brief Title: The Effect of Whole Blood Viscosity on Contrast-Induced Nephropathy Development in Patients Undergoing Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Professor Doctor, Bursa Postgraduate Hospital
Other Study IDs: YİEAH
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Percutaneous Coronary Intervention Patients
Keywords: Viscosity; Contrast; Nephropathy; Coronary Intervention
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood Viscosity Testing — we calculated WBV using the formula [(0.12 × hematocrit) + (0.17 × (total protein - 2.07)]. We defined CIN as the absolute (≥0.5 mg/dl) or relative increase (≥25%) in serum creatinine 48-72 h after exposure to a contrast agent compared with baseline serum creatinine values.

SUMMARY:
In our study, we aimed to investigate how whole blood viscosity (WBV) affects the development of contrast-induced nephropathy (CIN) in patients undergoing percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
In our study, 500 patients who applied to the cardiology clinic and underwent PCI for elective procedure, ST segment elevation myocardial infarction (STEMI), and non-STEMI were prospectively included. Before the procedure, we calculated WBV using the formula [(0.12 × hematocrit) + (0.17 × (total protein - 2.07)]. We defined CIN as the absolute (≥0.5 mg/dl) or relative increase (≥25%) in serum creatinine 48-72 h after exposure to a contrast agent compared with baseline serum creatinine values.

ELIGIBILITY:
Inclusion Criteria:

* patients between ages 18 and 90
* underwent PCI in our hospital between

Exclusion Criteria:

* Patients with chronic kidney disease (CKD) who underwent hemodialysis or peritoneal dialysis
* Patients who underwent to coronary bypass surgery within 48 h were excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study started with the approval of the local ethics committee. Five hundred patients between ages 18 and 90 who underwent PCI in our hospital between July 10, 2017, and October 31, 2017, were prospectively included. Informed consent forms were obtained from the patients. Patients with chronic kidney disease (CKD) who underwent hemodialysis or peritoneal dialysis for this reason and patients who underwent to coronary bypass surgery within 48 h were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Contrast Induced Nephropathy | 48 to 72 hours
  CIN was defined as an increase in serum creatinine levels greater than 0.5 mg/dl or 25% or more increase compared to basal serum creatinine levels 48 to 72 h after exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Hastanesi, Bursa, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camci S, Kinik M, Ari S, Ari H, Melek M, Bozat T. The predictive value of hemoglobin to creatinine ratio for contrast-induced nephropathy in percutaneous coronary interventions. Clin Chem Lab Med. 2022 Jun 22;60(9):1455-1462. doi: 10.1515/cclm-2022-0247. Print 2022 Aug 26. PMID 35727209
- [Derived] Kinik M, Camci S, Ari S, Ari H, Melek M, Bozat T. The effect of whole blood viscosity on contrast-induced nephropathy development in patients undergoing percutaneous coronary intervention. Postgrad Med. 2022 Jan;134(1):78-84. doi: 10.1080/00325481.2021.1997007. Epub 2021 Nov 10. PMID 34670475